CLINICAL TRIAL: NCT06729411
Title: Clinical Efficacy of a Novel Minimal Offloading Dressing for the Treatment of Plantar Diabetes-related Foot Ulcers: A Pilot Randomized Controlled Clinical Trial.
Brief Title: Minimal Offloading Dressing for the Treatment of Plantar Diabetes-related Foot Ulcers
Acronym: MOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Mateo López-Moral, DPM, PhD, Prof. Dr., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOD_2024
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer; Offloading
Keywords: diabetic foot; ulcer healing; offloading device; minimal offloading dressing; foot ulcer; healing
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group received minimal offloading dressing (MOD) treatments (Experimental): The MOD device was a monolayer device that can be applied directly to the participants skin via a non-irritative adhesive backing. The MOD was made of medium-density ethyl-vinyl acetate (40-45° Shore A hardness and 250-400-kg/cm2 density). The MOD is predesigned for three different locations: the first metatarsal head, central metatarsal heads, and fifth metatarsal. The MOD size ranged from size 35 to 48, which is measured according to the French system for each increase of 6.66 mm in length and 1.5 mm in width. All edges of the MOD were bevelled, and apertures were made to accommodate sites of plantar DFUs.
  Interventions: Device: Minimal Offloading dressing
- The control group received 15-mm felted foam treatments (Active Comparator): The felted padding used in the control group was made out of semi-compressed wool felt with an adhesive backing (Herbitas lab, 46134 Foios-Valencia, Spain). The padding thickness was 15 mm on the whole foot, and similar apertures to those used with the other offloading device were made to accommodate the sites of plantar ulceration.
  Interventions: Device: Felted foam

INTERVENTIONS:
Device: Minimal Offloading dressing — Metatarsal minimal offloading dressings (MODs) are standard offloading devices that are gaining attention. MODs offload a specific ulcerated area and could reduce variability when applying the device onto the skin. MODs are new predesigned devices that do not require any further adaptation or clinician skills and can be directly applied to an ulcerated metatarsal head using a non-irritating adhesive.
  Arms: The experimental group received minimal offloading dressing (MOD) treatments
Device: Felted foam — The felted padding used in the control group was made out of semi-compressed wool felt with an adhesive backing (Herbitas lab, 46134 Foios-Valencia, Spain). The padding thickness was 15 mm on the whole foot, and similar apertures to those used with the other offloading device were made to accommodate the sites of plantar ulceration.
  Arms: The control group received 15-mm felted foam treatments

SUMMARY:
A monocentre randomized controlled parallel (1:1) clinical trial was performed with consecutively selected individuals with diabetes and active diabetes-related foot ulcers (DFU). Participants were randomly assigned to control or treatment groups. The experimental group received MOD treatments, and the control group received 15-mm felted foam treatments. All participants wore a removable ankle-high offloading device.

Primary outcome measure was the 12-week healing rate. The time to healing was evaluated during a 12-week follow-up period. The secondary outcome measures included minor or major amputations related to the DFU during a follow-up period of 6 months.

DETAILED DESCRIPTION:
Participants and selection criteria Individuals who met the selection criteria were enrolled consecutively from our specialized outpatient diabetic foot unit. The inclusion criteria were confirmed type 1 or 2 diabetes mellitus, age >18 years, plantar DFU with Texas classification IA or IIA, glycaemic control confirmed by a haemoglobin A1c ≤ 10% (85.8 mmol/mol) in the previous 3 months, and a wound area of 1-30 cm2 at the time of inclusion. The exclusion criteria were critical limb ischaemia as defined by the Trans-Atlantic Inter-Society Consensus II guidelines, active DFU in the contralateral limb, major amputation (below or above the knee) of the contralateral limb, soft tissue infection, untreated diabetic foot osteomyelitis, or a need for walking aids. DFUs related to the lesser toes were excluded from the study due to the different indications for the offloading device.

Peripheral artery disease was confirmed by vascular assessment of the affected foot based on distal pedal pulse palpation, ankle-brachial index, toe brachial index, and transcutaneous oxygen pressure. Critical limb ischaemia was defined as an ankle-brachial index ≤ 0.4 and an ankle systolic blood pressure < 50 mm Hg or a toe systolic blood pressure < 30 mm Hg 13. The characteristics of DFUs were evaluated at baseline.

Interventions Participants were randomly assigned to control or treatment groups. After randomization, all participants were followed for 12 weeks to assess wound healing. Both groups received the same standard of care throughout the trial. The participants visited the outpatient clinic twice weekly, where the DFU was cleaned with sterile normal saline solution and debrided if needed. All wounds were dressed with neutral dressings, depending on the exudate level.

The experimental group received MOD treatments, and the control group received 15-mm felted foam treatments. All participants wore a removable ankle-high offloading device (Stabil-D device, Podartis s.r.l., Crocceta del Montello, Treviso, Italy) and a triple layer bandage to protect the foot shape. The surface of the wound area and photographs were assessed during each monthly visit until the wound healed or the end of the study. Planimetric wound-size measurements were performed by tracing the perimeter on an acetate grid with a fine-nibbed pen using Visitrak (Smith & Nephew, UK), and digital photographs were taken.

Minimal offloading dressing and felted padding The MOD device was a monolayer device that can be applied directly to the participants skin via a non-irritative adhesive backing. The MOD was made of medium-density ethyl-vinyl acetate (40-45° Shore A hardness and 250-400-kg/cm2 density). The MOD is predesigned for three different locations: the first metatarsal head, central metatarsal heads, and fifth metatarsal. The MOD size ranged from size 35 to 48, which is measured according to the French system for each increase of 6.66 mm in length and 1.5 mm in width. All edges of the MOD were bevelled, and apertures were made to accommodate sites of plantar DFUs.

The felted padding used in the control group was made out of semi-compressed wool felt with an adhesive backing (Herbitas lab, 46134 Foios-Valencia, Spain). The padding thickness was 15 mm on the whole foot, and similar apertures to those used with the other offloading device were made to accommodate the sites of plantar ulceration.

Outcome measures The primary outcome measure was the 12-week healing rate. Healing was defined as intact skin at the foot-ulcer site with complete epithelialization and no drainage. The time to healing was evaluated during a 12-week follow-up period. The secondary outcome measures included minor or major amputations related to the DFU during a follow-up period of 6 months. Delayed wound healing was defined as healing after the 12-week follow-up period. Transfer lesions were defined as a new ulcer located on the same foot secondary to an increase of pressure in areas adjacent to the primary DFU. Finally, adhesive irritation was defined as the presence of erythema and inflammation without the presence of a DFU secondary to contact with the offloading device.

Participants' health-related quality of life (HRQoL) was evaluated using the Diabetic Foot Ulcer Scale - Short Form (DFS-SF). The DFS-SF was applied in personal interviews that were conducted by a trained investigator (MLM). The DFS-SF contains 29 items based on six subscales: leisure, physical health, dependence/daily life, negative emotions, worry about ulcers/feet, and problems with ulcer care. Each item is rated on a 5-point Likert-type scale ranging from 1 ("not at all or none of the time") to 5 ("a great deal, all the time, or extremely"). Individual items on the instrument were reverse coded, and high scores on the DFS-SF indicate a high (good) HRQoL. The score of each subscale was calculated based on a scale of 0 (poorer HRQoL) to 100 (higher HRQoL). Each interview took approximately 15 min. The validated Spanish adaptation of the DFU-SF was used

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes mellitus.
* Age >18 years,
* Plantar DFU with Texas classification IA or IIA.
* Glycaemic control confirmed by a haemoglobin A1c ≤ 10% (85.8 mmol/mol) in the previous 3 months.
* Wound area of 1-30 cm2 at the time of inclusion.

Exclusion Criteria:

* Critical limb ischaemia as defined by the Trans-Atlantic Inter-Society Consensus II guidelines.
* Active DFU in the contralateral limb, major amputation (below or above the knee) of the contralateral limb.
* Soft tissue infection.
* Untreated diabetic foot osteomyelitis.
* Need for walking aids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Healing rate | 12-weeks
  Healing was defined as intact skin at the foot-ulcer site with complete epithelialization and no drainage

SECONDARY OUTCOMES:
Minor amputation | 6 months
  Any amputation below the ankle
Major amputation | 6 months
  Any foot amputation above de ankle, i.e below the knee amputation
Transfer lesions | 12-weeks
  Defined as a new ulcer located on the same foot secondary to an increase of pressure in areas adjacent to the primary DFU

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetic Foot Unit. Universidad Complutense de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will be shared if asked from any institution